CLINICAL TRIAL: NCT02921620
Title: A Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of PRX-102 on Gastrointestinal Symptoms in Naïve Fabry Disease Patients
Brief Title: Study to Evaluate the Safety and EffIcacy of PRX-102 on Gastrointestinal Symptoms in Naïve Fabry Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Protocol not feasible
Sponsor: Protalix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB-102-F10
Record Dates: First submitted 2016-09-26; First posted 2016-10-03 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Fabry Disease
Keywords: Gastrointestinal symptoms; Diarrhea; Abdominal pain
MeSH Terms: conditions — Fabry Disease; Diarrhea; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PRX-102 (Experimental): PRX-102 infusions every 2 weeks
  Interventions: Biological: PRX-102
- Placebo (Placebo Comparator): Placebo infusions every 2 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PRX-102 — Intravenous
  Other Names: pegunigalsidase alfa; recombinant human alpha galactosidase-A
  Arms: PRX-102
Other: Placebo — Intravenous
  Arms: Placebo

SUMMARY:
The study will be a randomized, double blind, placebo-controlled study of the safety and efficacy of PRX-102 in ERT naïve male patients randomized 1:1. Patient age will be 14 to 45 years. Patients must have diarrhea defined as ≥ 3 stools a day with an average consistency of ≥ 5.5 on the Bristol Stool Form Scale (BSFS) by patient electronic diary and moderate to severe gastrointestinal symptoms as defined by the Irritable Bowel Symptom Severity Score (IBSSS) Part 1 average > 175 derived from at least two IBSSS assessments during screening period. Patients will receive intravenous infusions of PRX-102 1 mg/kg or placebo every two weeks for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 14-45 years, naïve to enzyme replacement therapy (ERT) or off ERT or off chaperone treatment for at least 6 months and negative for anti-PRX-102 antibodies
* A documented diagnosis of Fabry disease: Plasma and/or leucocyte alpha galactosidase activity (by activity assay) less than lower limit of normal (LLN)
* eGFR by CKD-EPI > 30 ml/min/1.73 m2
* Moderate to severe gastrointestinal symptoms as defined by:

  * Average score of > 175 from at least two Irritable Bowel Symptom Severity Score (IBSSS) Part 1 assessments before randomization.
  * Average stool consistency of ≥ 5.5 on the Bristol Stool Form Scale (BSFS) by patient diary during 2 weeks prior to randomization out of the 4 week of screening period and
  * ≥ 3 stools a day with a consistency of ≥ 5 on the BSFS during the week before randomization.
* Completed electronic BSFS diary on at least 6 of the 7 days during the week prior to randomization AND at least 11 of the 14 days during the 2 weeks prior to randomization.

Exclusion Criteria:

* Patients will be evaluated to rule out other gastrointestinal comorbidity than Fabry disease as responsible for the gastrointestinal symptoms by:

  i. Medical History for non Fabry gastrointestinal comorbidity ii. Occult blood in stool iii. Stool culture for bacteria and parasites iv. Calprotectin in stool v. Sigmoidoscopy
* Use of any kind of laxatives
* Initiation of anti-diarrheal medications during the screening period
* History of renal dialysis or transplantation
* Use of, or change in dose of, angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) for less than 4 weeks prior to screening
* Cardiovascular event (myocardial infarction, unstable angina) in the 6 month period before randomization
* Congestive heart failure NYHA Class IV
* Cerebrovascular event (stroke, transient ischemic attack) in the 6 month period before randomization
* Known history of hypersensitivity to Gadolinium contrast agent
* Known allergies to ERT
* Presence of any medical, emotional, behavioral or psychological condition that, in the judgment of the Investigator and/or Medical Director, would interfere with the patient's compliance with the requirements of the study

Ages: 14 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
IBSSS Part 1 | Every 2 weeks for 6 months
  Irritable Bowel Syndrome Severity Score

SECONDARY OUTCOMES:
Stool frequency | After every bowel movement for 6 months
  from BSFS diary
Body Weight | Every 2 weeks for 6 months
Plasma Lyso-Gb3 | Every 4 weeks for 6 months
Plasma Gb3 | Every 4 weeks for 6 months
Urine Lyso-GB3 | Every 6 weeks for 6 months
Frequency of pain medication use | Every 2 weeks for 6 months

OTHER OUTCOMES:
Anti-PRX-102 antibodies | Every 4 weeks for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raul Chertkoff, MD, Study Director — Protalix Ltd.

IPD SHARING:
Plan to Share IPD: Undecided